### INFORMED CONSENT FORM FOR ONLINE SURVEY

**To learn more** about the study or see the questions in the survey, please visit <a href="https://safe-firearm.org/parent-survey/henry-ford-health/">https://safe-firearm.org/parent-survey/henry-ford-health/</a>.

#### TITLE OF THE RESEARCH STUDY:

A comparative effectiveness trial of strategies to implement firearm safety promotion as a universal suicide prevention strategy in pediatric primary care

# PRINCIPAL INVESTIGATOR & EMERGENCY CONTACT: [REMOVED]

**INTRODUCTION**: You are invited to participate in this research study because your child recently attended a well-visit at Henry Ford Health (HFH). You are being invited to participate in a survey about topics that may have been discussed at your child's visit. The survey can be completed online on REDCap, over the phone, or via a mailed survey. The purpose of this survey is to help us understand whether firearms are discussed during well-visits and how parents perceive these discussions. It will take approximately 1-3 minutes to complete the survey. We may also contact you in the future to ask if you are interested in participating in additional activities related to this research.

To qualify for the study, you must be 18 years of age or older. You also must be a parent and/or legal guardian of a child age 5-17 who attended a well-visit recently at a participating HFH clinic. Lastly, you must be a resident of the United States and speak English.

This research study is funded by the National Institute of Mental Health.

**PARTICIPATION**: Your participation in this survey is voluntary. You may refuse to take part in the research, skip specific questions, or exit the survey at any time without penalty. Your doctor will not be upset with your decision. If you decide to participate, your doctor will not be able to see your survey responses. If you decide you do not want your responses used, you can submit a written request to the research team to no longer use your survey responses and we will then destroy your responses.

**BENEFITS**: You will receive no direct benefits from participating in this research study. However, you may find satisfaction in sharing your thoughts on your experience at your recent well-visit.

**COMPENSATION**: After completing this survey, you will be entered into a drawing to receive a \$100 gift card. We will distribute 150 gift cards at HFH over the two and a half years of the study. You will only be eligible to be entered into the drawing if you meet the eligibility criteria described above. The compensation will be in the form of a ClinCard, which is a specially designed debit card for clinical research that works like a bank debit card. The ClinCard is administered by an outside company, which will use your information only to pay you. Your information will not be used for any other purposes and will not be given or sold to any other company. All information is stored in a secure fashion and will be deleted from our records once the study has been completed and the funds on your ClinCard have been exhausted.

You may use this card at any store that accepts credit cards. You may also withdraw cash. Please be aware that there may be fees drawn against the balance of the card for cash withdrawals and inactivity. You will receive additional information on how you can use this card and any fees that may apply. If you receive \$600 or more for taking part in this research study or a combination of studies in one tax year, you will be sent a 1099 form for tax purposes.

**RISKS**: The possible risks of participating in this study include possible discomfort that may arise from completing the survey and loss of confidentiality, or that someone outside of the study will see your information.

**CONFIDENTIALITY**: All responses will be treated confidentially. We have taken steps to protect your responses. The information obtained in this survey will only be used for this project. Only authorized people on the research team and the University of Pennsylvania Institutional Review Board will have access to the information. In reports, your answers will be grouped with those of others. All data reported through REDCap, our web-based, HIPAA-compliant survey platform, will be secured using HIPAA-compliant technology and all data will be maintained on a HIPAA-compliant server.

**FUTURE USE:** In addition to the data used as described above, we will also store your de-identified data for future use. De-identified means that all identifiers have been removed. The information may be shared with other researchers within Penn, or other research institutions, or the National Institutes of Health. It would not be possible for future researchers to identify you as we would not share any identifiable information about you with future researchers. This can be done without again seeking your consent in the future, as permitted by law. The future use of your information only applies to the information collected on this study.

**CONTACT**: If you have questions at any time about the study or the procedures, you may contact [PRINCIPAL INVESTIGATORS @ CONTACT INFORMATION]. If you have any questions about your rights as a human research participant at any time before, during, or after participation, please contact the University of Pennsylvania Institutional Review Board (IRB) at (215) 898-2614 or the Henry Ford Health IRB Administration Office by phone at (313) 874-4464 or by email at research\_admin@hfhs.org.

**ELECTRONIC CONSENT**: Please select your choice below. You may print a copy of this consent form for your records. Clicking on the "Agree" button indicates that:

- You have read the above information
- You voluntarily agree to participate
- You are 18 years of age or older
- You are the parent or guardian of the child and you took the child to the well-child visit

If you are not the parent or legal guardian who attended the recent well-child visit with your child, please close this consent form and forward the survey invitation message to the parent or legal guardian who attended the well-child visit. If a parent or legal guardian did not attend the well-child visit, please close out and disregard this survey.

| □ Agree |
|---|
| □ Disagree |
| ** FOR RESEARCH TEAM ONLY ** |
| If verbal consent was obtained from the parent/legal guardian over the phone, please complete the following: |
| Name of parent/guardian from whom consent was obtained: |
| Print name of person who obtained consent: |
| Signature of person who obtained consent: |
| Date: |

#### INFORMED CONSENT FORM FOR ONLINE SURVEY

**To learn more** about the study or see the questions in the survey, please visit <a href="https://safe-firearm.org/parent-survey/kaiser-permanente-colorado/">https://safe-firearm.org/parent-survey/kaiser-permanente-colorado/</a>.

### TITLE OF THE RESEARCH STUDY:

A comparative effectiveness trial of strategies to implement firearm safety promotion as a universal suicide prevention strategy in pediatric primary care

## PRINCIPAL INVESTIGATOR & EMERGENCY CONTACT: [REMOVED]

**INTRODUCTION**: You are invited to participate in this research study because your child recently attended a well-visit at Kaiser Permanente Colorado (KPCO). You are being invited to participate in a survey about topics that may have been discussed at your child's visit. The survey can be completed online on REDCap, over the phone, or via a mailed survey. The purpose of this survey is to help us understand whether firearms are discussed during well-visits and how parents perceive these discussions. It will take approximately 1-3 minutes to complete the survey. We may also contact you in the future to ask if you are interested in participating in additional activities related to this research.

To qualify for the study, you must be 18 years of age or older. You also must be a parent and/or legal guardian of a child age 5-17 who attended a well-visit recently at a participating KPCO clinic.

This research study is funded by the National Institute of Mental Health.

**PARTICIPATION**: Your participation in this survey is voluntary. You may refuse to take part in the research, skip specific questions, or exit the survey at any time without penalty. Your doctor will not be upset with your decision. If you decide to participate, your doctor will not be able to see your survey responses. If you decide you do not want your responses used, you can submit a written request to the research team to no longer use your survey responses and we will then destroy your responses.

**BENEFITS**: You will receive no direct benefits from participating in this research study. However, you may find satisfaction in sharing your thoughts on your experience at your recent well-visit.

**COMPENSATION**: After completing this survey, you will be entered into a drawing to receive a \$100 gift card. We will distribute 150 gift cards at KPCO over the two and a half years of the study. You will only be eligible to be entered into the drawing if you meet the eligibility criteria described above. The compensation will be in the form of an electronic gift card (e.g., Amazon.com).

**RISKS**: The possible risks of participating in this study include possible discomfort that may arise from completing the survey and loss of confidentiality, or that someone outside of the study will see your information.

**CONFIDENTIALITY**: All responses will be treated confidentially. We have taken steps to protect your responses. The information obtained in this survey will only be used for this project. Only authorized people on the research team and the University of Pennsylvania Institutional Review Board will have access to the information. In reports, your answers will be grouped with those of others. All data reported through REDCap, our web-based, HIPAA-compliant survey platform, will be secured using HIPAA-compliant technology and all data will be maintained on a HIPAA-compliant server.

**FUTURE USE:** In addition to the data used as described above, we will also store your de-identified data for future use. De-identified means that all identifiers have been removed. The information may

be shared with other researchers within Penn, or other research institutions, or the National Institutes of Health. It would not be possible for future researchers to identify you as we would not share any identifiable information about you with future researchers. This can be done without again seeking your consent in the future, as permitted by law. The future use of your information only applies to the information collected on this study.

**CONTACT**: If you have questions at any time about the study or the procedures, you may contact [PRINCIPAL INVESTIGATORS @ CONTACT INFORMATION]. If you have any questions about your rights as a human research participant at any time before, during, or after participation, please contact the University of Pennsylvania Institutional Review Board (IRB) at (215) 898-2614.

**ELECTRONIC CONSENT**: Please select your choice below. You may print a copy of this consent form for your records. Clicking on the "Agree" button indicates that:

- You have read the above information
- You voluntarily agree to participate
- You are 18 years of age or older
- You are the parent or guardian of the child and you took the child to the well-child visit

If you are not the parent or legal guardian who attended the recent well-child visit with your child, please close this consent form and forward the survey invitation message to the parent or legal guardian who attended the well-child visit. If a parent or legal guardian did not attend the well-child visit, please close out and disregard this survey.

| □ Agree |
|---|
| □ Disagree |
| ** FOR RESEARCH TEAM ONLY ** |
| If verbal consent was obtained from the parent/legal guardian over the phone, please complete the following: |
| Name of parent/guardian from whom consent was obtained: |
| Print name of person who obtained consent: |
| Signature of person who obtained consent: |
| Date: |

### INFORMED CONSENT FORM FOR WEB SURVEY

**TITLE OF THE RESEARCH STUDY:** A comparative effectiveness trial of strategies to implement firearm safety promotion as a universal suicide prevention strategy in pediatric primary care

# PRINCIPAL INVESTIGATORS & EMERGENCY CONTACTS: [REMOVED]

You are invited to participate in a survey about your clinic and your opinions and experiences around discussing firearm safety with patients. You may be asked questions about the *S.A.F.E. Firearm* program, firearms, suicide prevention, your experiences, demographics, and/or characteristics of the clinic(s) that you work in. This is a research project being conducted by Dr. Rinad Beidas at Northwestern University, Dr. Kristin Linn at the University of Pennsylvania, Dr. Brian Ahmedani at Henry Ford Health, and Dr. Jennifer Boggs at Kaiser Permanente Colorado. It should take approximately 15 minutes to complete this survey. If you have any questions about your rights as a human research participant, please contact the University of Pennsylvania Institutional Review Board (IRB) at 215-898-2614.

### PARTICIPATION:

You are being asked to join this study because you are a clinician or leader in a pediatrics or family medicine clinic at Kaiser Permanente Colorado or Henry Ford Health.

Your participation in this survey is voluntary. You may refuse to take part in the research or exit the survey at any time without penalty. You are free to decline to answer any particular question you do not wish to answer for any reason.

If you decide to participate, you will navigate to the next page of this survey and you will be asked to answer several questions. Your participation in this survey will involve you answering questions that will help us understand you and your clinic, including your opinions and experiences around the *S.A.F.E. Firearm* program and suicide prevention, your personal experiences with firearms, and characteristics of the clinic(s) that you work in.

**BENEFITS**: You will receive no direct benefits from participating in this research study. However, your participation could help us understand clinicians' and leaders' experiences and opinions around discussing firearm safety and delivering the *S.A.F.E. Firearm* program to their patients.

**COMPENSATION:** If allowed by your health system, you will receive a \$20 e-gift card for participating in this survey or a \$20 altruistic gift will be made on your behalf to a suicide prevention charity.

Version 12/13/2022 

**RISKS**: The only possible risk of participating in this study is the potential for breach of confidentiality.

**CONFIDENTIALITY**: We have taken steps to protect your confidentiality. Only authorized people on the research team and the University of Pennsylvania Institutional Review Board will have access to the information. In reports, your answers will be grouped with those of others. We will never mention your name. With all of these safeguards, it is still possible that your confidentiality may be compromised.

We will maintain your confidentiality by ensuring that:

- Information will only be used and shared with those involved in this research study.
- All data reported through the HIPAA-compliant survey platform (called REDCap) will be used by the research team in compliance with all applicable laws and regulations.
- All data will be stored on HIPAA-compliant platforms maintained by the University of Pennsylvania Perelman School of Medicine and Northwestern University.
- Files kept on the computer will not contain identifying information such as your name, email address, or any other personal identifiable information (PII).

### WHAT MAY HAPPEN TO YOUR INFORMATION COLLECTED DURING THIS

**STUDY**: Your information will be de-identified. De-identified means that all identifiers have been removed. The information could be stored and shared for future research in this de-identified fashion. Your survey responses will **not** be shared with anyone from your health system in an identified fashion. The de-identified information may be shared with other researchers within Penn or Northwestern, or other research institutions, or the National Institutes of Health. It would not be possible for future researchers to identify you as we would not share any identifiable information about you with future researchers. This can be done without again seeking your consent in the future, as permitted by law. The future use of your information only applies to the information collected on this study.

**CONTACT**: If you have questions at any time about the study or procedures, you may contact the principal investigators listed at the top of this consent form.

If you feel you have **not** been treated according to the descriptions in this form, or that your rights as a participant in research have not been honored during the course of this project, or you have any questions, concerns, or complaints that you wish to address to someone other than the investigators, you can call the University of Pennsylvania Institutional Review Board at 215-898-2614.

**ELECTRONIC CONSENT:** Please select your choice below. You may print a copy of this consent form for your records. Clicking on the "Agree" button indicates that:

- You have read the above information
- You voluntarily agree to participate

Version 12/13/2022 

| • | You are 18 years of age or older |
|---|----------------------------------|
| | Agree |
| | Disagree |

Version 12/13/2022 